CLINICAL TRIAL: NCT05359133
Title: A Randomized, Double-Blind, Placebo Controlled, Multicenter, Efficacy and Safety Trial of Single Cycle Tetrodotoxin in the Treatment of Chemotherapy Induced Neuropathic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to lack of funding to continue the study.
Sponsor: Wex Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTX-CINP-202
Record Dates: First submitted 2022-04-25; First posted 2022-05-03 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-08

CONDITIONS: Chemotherapy-induced Neuropathic Pain; Chemotherapy-induced Peripheral Neuropathy
Keywords: CINP; Chemotherapy-induced Neuropathic Pain; Pain; Neuropathy
MeSH Terms: conditions — Pain | interventions — Tetrodotoxin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tetrodotoxin for injection (Active Comparator): 30 µg, 1 ml SC injection in the thigh or abdomen, twice daily for 4 Days
  Interventions: Drug: Tetrodotoxin
- Placebo (Placebo Comparator): 1.0 mL of placebo, SC injection in the thigh or abdomen, twice daily for 4 Days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetrodotoxin — TTX for Injection, 30 µg/mL, is a sterile, nonpyrogenic, white, lyophilized powder provided in a 5 mL glass single-use vial with a rubber stopper and aluminum overseal. Upon reconstitution of the lyophilized product with 1.1 mL of sterile water for injection, each vial delivers 1 mL of fluid containing 30 µg of TTX with a pH of 4.0 to 5.5
  Other Names: Halneuron
  Arms: Tetrodotoxin for injection
Drug: Placebo — Placebo for injection is a sterile 0.9% sodium chloride injection or normal saline for injection. To ensure blinding, subjects receiving placebo will receive the same volume (1.0 mL) for injection to match the volume used for the cohorts assigned to receive active trial drug.
  Route and frequency: 1.0 mL of placebo, SC injection in the thigh or abdomen, twice daily for 4 Days in each treatment Cycle.
  Other Names: Sterile 0.9% sodium chloride injection
  Arms: Placebo

SUMMARY:
To be eligible for the trial, subjects must have ongoing moderate to severe neuropathic pain related to a prior course of platinum and/or taxane chemotherapy and have no clinical evidence of actively progressive disease.

The trial period will comprise a Screening period (up to 35 Days), randomization and a 4-day treatment period, followed by a 12-week follow up period (12 weeks total after initial treatment), and an End-of-Trial/Follow-up visit which will occur at Week 13. This is a study to research the effects of the study drug on neuropathic pain compared placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥21 years.
* Subjects and their partners must agree to using effective methods of birth control from the time of signature of the informed consent form up until 30 days following the end of the Treatment Period.
* Subjects with neuropathic pain attributed to platinum and/or taxane chemotherapy for a minimum of 3 months duration from screening.
* Subjects with cancer who have completed a chemotherapy regimen that included taxanes or platinums (or in combination) and have no clinical evidence of actively progressive disease. Subjects must have undergone at least a 90-Day washout period between the last dose of cytotoxic chemotherapy/radiotherapy agent and randomization. Concurrent hormonal therapy and immunotherapy that do not cause neuropathy are permitted.
* Subjects with a score of 4 or higher out of 10 on the Diagnosing Neuropathic Pain-DN4 Questionnaire (Appendix F) at Screening.
* Subjects must have at least 10 non-missing scores in the 14 Days prior to randomization during their Baseline Period.
* Subjects with moderate to severe neuropathic pain that has been stable for 14 Days. Stable pain will be confirmed using an 11-point (0-10) NPRS. To establish moderate or severe stable pain, the average daily pain scores during the 14-Day Baseline Period must be ≥4 with fluctuation in the daily pain score of ≤2 points in increase or decrease. Subjects with an average pain score >9 at Baseline will be excluded.
* Subjects with an Eastern Cooperative Oncology Group Performance Status score of 0 or 1 (Oken et al, 1982).
* Subjects who are able to communicate well with the trial staff and to comply with the trial requirements (restrictions, appointments, and examination schedule).
* Subjects who are able to complete the trial-related questionnaires independently in either English or in the local language.
* Subjects who sign an informed consent document (prior to the performance of any trial related procedures).

Exclusion Criteria:

* History of peripheral neuropathy attributed to any cause other than platinum or taxane chemotherapy (e.g., radiotherapy, vinca alkaloids, diabetes, alcohol, toxin, hereditary, human immunodeficiency virus, or severe malnutrition).
* Subjects who have received TTX at any time prior to enrolment.
* Subjects receiving agents known to cause peripheral neuropathy within 90 Days of randomization.
* Current use of any other therapy (including alternative nonmedical therapy) for the treatment of neuropathic pain within 60 Days of randomization unless the dose is stable for the 60 Days immediately prior to randomization. Subjects who fail this criterion can be rescreened after 60 Days of stability.
* Current use of opioids or plans to start using opioids during the study period. However, opioids at doses of ≤90 mg morphine equivalents per day are permitted as long as subject is on stable dose for at least 60 days prior to randomization and plan on staying on that stable dose (fixed dose and schedule) throughout the study.
* Subjects who require rescue medication for breakthrough pain with medication other than acetaminophen or Ibuprofen. Before and after randomization, acetaminophen will be allowed at doses up to 2600 mg per day <3 times a week or Ibuprofen will be allowed at doses up to 1200 mg per day <3 times a week.
* Any concomitant medication that prolongs the QT or QRS interval unless on a stable dose for 60 Days prior to randomization.
* Subjects with known impaired renal function as determined by a screening serum creatinine >1.5x normal.
* Subjects who have not recovered from all toxicities related to chemotherapy to < grade 1 or mild AE's with the exception of CINP.
* Subjects who have inadequate organ function tests including: Hgb < 10 g/dl; ANC < 1500/µL; Plt. count < 100,000/µL; liver function (ALT and/or AST) more than 2 times the upper limit of normal.
* Subjects with urinary retention.
* Subjects with documented bone metastases at the time of trial entry.
* Subjects with predicted life expectancy of <8 months.
* Subjects scheduled for chemotherapy or radiotherapy between Screening and the End of Trial visit (Week 13).
* Current use of lidocaine (including Lidoderm) and other types of sodium channel antiarrhythmic drugs within 30 Days of randomization.
* Subjects who have been injected with Botulinum toxin (e.g., Botox®) in the 3 months prior to randomization, or who plan to receive a Botulinum toxin injection during the study period.
* Subjects who require regular antiemetic medication.
* Current use of tricyclic antidepressant medication, anticonvulsants, or monoamine oxidase inhibitors. Stable use of those medications for at least 2 months is permissible if the subject has qualifying pain and plans to remain on a stable dose throughout the trial.
* Subjects will be excluded if they have a current diagnosis of uncontrolled Major Depressive Disorder.
* Subjects with current uncontrolled asthma, carbon dioxide retention, or oxygen saturation <92% on room air, or require oxygen therapy at any concentration.
* Subjects with second- or third-degree heart block or prolonged QTc interval (corrected for rate) on screening electrocardiogram (ECG) (i.e., confirmed >450 msec for men and >470 msec for women on repeated occasion) or any other active cardiac arrhythmia or abnormality that might constitute a clinical risk.
* Subjects with neuromuscular conditions, including but not limited to any impairment that influence swallowing or breathing function.
* Use of an investigational agent within 30 Days prior to Screening or scheduled to receive an investigational drug other than TTX during the course of the trial.
* History of alcoholism, or current intake deemed excessive by the investigator or routine use averaging >3 units of alcohol per day.
* Active substance abuse or drug dependency in the opinion of the investigator, including prescription drug abuse.
* Women who are pregnant or breast feeding.
* Any other condition that in the opinion of the investigators is likely to interfere with treatment, impede data collection, or that poses a risk to the subject.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
NPRS Pain reduction - at week 4 | At week 4
  The Change from Baseline (average of Days -14 to -1) at Week 4 in average weekly NPRS scores in subjects treated with TTX compared to Placebo

SECONDARY OUTCOMES:
NPRS Pain reduction - at week 8 | At week 8
  The Change from Baseline (average of Days -14 to -1) at Week 8 in average weekly NPRS scores in subjects treated with TTX compared to Placebo
NPRS Pain reduction - at week 12 | At week 12
  The Change from Baseline (average of Days -14 to -1) at Week 12 in average weekly NPRS scores in subjects treated with TTX compared to Placebo

OTHER OUTCOMES:
AUC up to week 12 | baseline to week 12
  AUC calculated on the Change from Baseline through Week 12 in weekly average NPRS scores.
NPRS Pain reduction - weekly | baseline to week 12
  Change from Baseline to each study week through Week 12 in Average Weekly NPRS scores
NPRS Pain reduction - weekly | baseline to week 12
  Percent Change from Baseline to each study week through Week 12 in Average Weekly NPRS scores
Subjects with at least 30% reduction in pain | baseline to week 12 (assessed weekly)
  Proportion of responders at Week 12, defined as subjects showing a 30% or greater reduction from overall Baseline (Week -1 & week -2) to Week 12 in weekly average NPRS score.
Subjects with at least 50% reduction in pain | baseline to week 12 (assessed weekly)
  Proportion of responders at Week 12, defined as subjects showing a 30% or greater reduction from overall Baseline (Week -1 & week -2) to Week 12 in weekly average NPRS score.
Time to response | Day 1 to week 12
  Time to first response defined as (30%/50%) reduction from overall Baseline in weekly average NPRS score
Duration of response | Day 1 to week 12
  Duration of response defined as time from initial (30%/50%) reduction from overall baseline in weekly average NPRS score to first loss of response.
BPI change | Baseline to Week 12
  Change from Baseline to each study visit through Week 12 in quality of life and pain intensity measures using the Brief Pain Inventory (BPI).
NPSI change | Baseline to Week 12
  Change from Baseline to each study visit through Week 12 in neuropathic pain symptoms using the Neuropathic Pain Symptoms Inventory (NPSI)
POMS change | Baseline to Week 12
  Change from Baseline to each study visit through Week 12 in Profile of Mood States (POMS2) total mood disturbance, and each of the 6 specific subscales.
Percent of subjects taking Rescue Medication | Baseline to Week 12
  Percentage of subjects taking allowed and prohibited rescue medication at each week, including Week 12.
Average rescue medication consumed | Baseline to Week 12
  Average per-subject consumption of allowed and prohibited rescue medication at each week, including Week 12
Patient global impression of change questionnaire | at week 12
  Subjects' Global Impression of Change responses at each visit through the End-of-Trial visit.
Proportion of responders (30%/50%) | weekly until week 12
  Proportion of responders (30%/50%) at each study week through Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Walter Korz, Study Director — COO
Locations (15):
- United States (15):
  - Syrentis Clinical Research, Santa Ana, California
  - Providence Medical Foundation, Santa Rosa, California
  - MEDSOL Clinical Research Center, Port Charlotte, Florida
  - Care Access Research, Macon, Georgia
  - Paradigm Clinical Research, Boise, Idaho
  - Clinical Trials of SWLA, Lake Charles, Louisiana
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - St Luke's Hospital of Kansas City, Kansas City, Missouri
  - Care Access Research, Clifton, New Jersey
  - ES Clinical Research Group, Garden City, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Oklahoma Cancer Specialists and Research Institute (OCSRI), Tulsa, Oklahoma
  - Center for Oncology and Blood Disorders (COBD), Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas